CLINICAL TRIAL: NCT02945631
Title: Quarterback 22: A Phase II Clinical Trial of Sequential Therapy and De-Intensified Chemoradiotherapy for Locally Advanced HPV Positive Oropharynx Cancer
Brief Title: Quarterback 2b - Sequential Therapy With Reduced Dose Chemoradiotherapy for HPV Oropharynx Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Marshall Posner, MD, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-0609
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2024-07-05 (Actual); Status verified 2024-03

CONDITIONS: Locally Advanced HPV Positive Oropharynx Cancer
Keywords: HPV; Induction Chemotherapy; De-Intensified Chemoradiotherapy; Oropharynx Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: Yes

ARMS (1):
- Reduced Dose Radiation (Experimental): All patients will receive daily radiation treatment with intensity-modulated radiotherapy (IMRT) - PTV56 and PTV50.4. Treatment will be given 5 days per week and will not routinely be delivered on Saturday, Sunday or major holidays unless a treatment is missed during the week due to technical and/or medical reasons. No more than 5 treatments should be given per week.
  Interventions: Radiation: PTV56; Radiation: PTV50.4

INTERVENTIONS:
Radiation: PTV56 — total dose of 56 Gy in 2.0 Gy/fraction x 28 fractions.
Radiation: PTV50.4 — total dose of 50.4 Gy in 1.8 Gy /fraction x 28 fractions.

SUMMARY:
The purpose of this study is to establish the efficacy and toxicity of low dose chemoradiotherapy after induction chemotherapy in patients with locally advanced HPV+ oropharynx cancer and establish prognostic factors that would apply to help select patients for this treatment in the future.

DETAILED DESCRIPTION:
In general, patients with Human Papilloma Virus Oropharynx Cancer (HPVOPC) are young and will live for prolonged periods. They are at high risk for long-term toxicity and mortality from radiotherapy. While the long-term consequences of chemotherapy for head and neck cancer are relatively constrained, high-dose radiotherapy (RT) and chemoradiotherapy (CRT) substantially impact on local tissues and organ function and result in a significant rate of late mortality and morbidity in patients. Studies are now being designed to reduce the impact of RT and CRT for patients. Identifying appropriate endpoints and study arms which will allow an early assessment of outcomes will be problematic, particularly for equivalence studies wherein survival differences are small, and where prolonged time periods and large patient numbers are necessary to accurately assess outcomes. For Sequential Therapy as given with TAX 324, 3-year PFS may be an appropriate endpoint. The same may not be possible for CRT. The best example of changing outcomes in CRT trials would be R91-11, in which a premature negative conclusion regarding the efficacy of induction therapy was published with the early analysis. Late toxicity and morbidity, a hallmark of upfront cisplatin-based CRT trials, led to equivalence between induction therapy and CRT for laryngectomy-free survival at 5 years, and more importantly a non-significant relative 10% improvement in overall survival in the PF induction arm compared to the CRT arm which included an every 3-week bolus cisplatin for 3 cycles during radiotherapy.

The survival results in HPVOPC achieved in TAX 324 and preliminary data from ECOG 1308 strongly suggest that it might be possible to reduce long-term morbidity in HPVOPC and preserve survival perhaps by better patient selection and by reducing radiotherapy intensity in the context of ST for more advanced cases. Best approach of HPV-negative disease might be with novel therapies and more aggressive Sequential Therapy (ST) or CRT.

Current radiation dose reduction trials are under way in ECOG, RTOG and other radiation based groups. The data from TAX 324 suggest that it is possible to reduce the radiation dose because of the superior progression free survival and the ability to select risk based CRT.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria to be eligible to participate in the study. Patients may enroll in the study if they meet all of the entry criteria, were candidates for induction chemotherapy regardless of HPV status and have to start therapy for logistic reasons prior to p16 and HPV testing. They will enter the experimental post-Induction portion of the study if the surgical specimens or biopsies are proven to be HPV+ on PCR testing. Patients who are HPV negative will be taken off study and treated with SOC radiotherapy and surgery:

* Participants must have histologically or cytologically confirmed squamous cell carcinoma of the oropharynx, hypopharynx, supraglottic larynx, nasal cavity, unknown primary, or nasopharynx that is p16 and HPV positive. Tissue from the primary site or lymph node must be available for biomarker studies and for PCR testing. IHC must be performed in a lab verified by the central laboratory or the slides must be available for review by the central laboratory and PCR must be done in the central laboratory prior to radiotherapy. HPVPCR must be performed and results available for reduced dose therapy after induction.
* Patients who are on the Quarterback Trial when Quarterback 2 is activated and who have been randomized to radiotherapy arm will be asked to transfer to this trial and receive the Quarterback 2 defined radiotherapy.
* Stage 3 or 4 disease without evidence of distant metastases.
* At least one clinically evaluable or uni- or bi-dimensionally measurable lesion by RECIST 1.1 criteria.
* Age ≥ 18 years.
* No previous surgery, radiation therapy or chemotherapy for SSCHN (other than biopsy or tonsillectomy) is allowed at time of study entry.
* ECOG performance status of 0 or 1.
* No active alcohol addiction (as assessed by medical caregiver and defined as at least 6 months without activity).
* Participants must have adequate bone marrow, hepatic and renal functions as defined below:
* - Hematology:
* - Neutrophil count ≥ 1.5 x 10^9/l.
* - Platelet count ≥ 100 x 10^9/l.
* - Hemoglobin ≥ 10g/dl.
* - Renal function ≥ 60 ml/min (actual or calculated by the Cockcroft-Gault method) as follows: CrCl (ml/min) = (140-age)(weight kg)/(mL/min) / 72 x serum creatinine (mg/dL)
* - N.B. For females, use 85% of calculated CrCl value. Or a Creatinine ≤ the upper limits of normal
* - Hepatic:
* - Total Bilirubin ≤ institutional upper level of normal (ULN)
* - AST or ALT and Alkaline Phosphatase must be within the range allowing for eligibility
* Women of childbearing potential must have a negative pregnancy test within 7 days of starting treatment.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients with Gilbert's Disease and absent hepatic pathology by history and clinical assessment may be treated on study with bilirubin > the ULN for the institution if other liver functions studies are within the normal range

Exclusion Criteria:

* Pregnant or breast feeding women, or women and men of childbearing potential not willing to use adequate contraception while on treatment and for at least 3 months thereafter.
* Previous or current malignancies at other sites, with the exception of adequately treated in situ carcinoma of the cervix, basal or squamous cell carcinoma of the skin, thyroid cancer, or other cancer curatively treated by surgery and with no current evidence of disease for at least 5 years.
* Symptomatic peripheral neuropathy grade > 2 by NCI Common Terminology Criteria (NCI-CTC) version 4.
* Symptomatic altered hearing > grade 2 by NCI-CTCv4 criteria.These patients can be entered by substituting carboplatin for cisplatin with an AUC of 6.0
* Other serious illnesses or medical conditions including but not limited to:
* - Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
* - History of significant neurologic or psychiatric disorders including dementia or seizures
* - Active clinically significant uncontrolled infection
* - Active peptic ulcer disease defined as unhealed or clinically active
* - Hypercalcemia
* - Active drug addiction including alcohol, cocaine or intravenous drug use defined as occurring within the 6 months preceding diagnosis
* - Chronic Obstructive Pulmonary Disease, defined as being associated with a hospitalization for pneumonia or respiratory decompensation within 12 months of diagnosis. This does not include obstruction from tumor
* - Autoimmune disease requiring therapy, prior organ transplant, or HIV infection
* - Interstitial lung disease
* - Hepatitis C by history, and confirmed by serology
* Patients that have experienced an involuntary weight loss of more than 25% of their body weight in the 2 months preceding study entry.
* Concurrent treatment with any other anticancer therapy.
* Participation in an investigational therapeutic drug trial within 30 days of study entry.
* Active smoking or a cumulative pack year history of > 20 pack years, active smoking is (Defined as ≥ 1 cigarette per day) within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 3 years
  The comparative rate of progression free survival
Progression Free Survival | 5 years
  The comparative rate of progression free survival

SECONDARY OUTCOMES:
Local-regional control (LRC) | 3 years
  The comparative rate of local-regional control
Local-regional control (LRC) | 5 years
  The comparative rate of local-regional control
Overall Survival (OS) | 3 years
Overall Survival (OS) | 5 years
Acute Toxicity | 5 years
  Rate of acute toxicity
Long Term Toxicity | 5 years
  Rate of long term toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Posner, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaturvedi AK, Engels EA, Pfeiffer RM, Hernandez BY, Xiao W, Kim E, Jiang B, Goodman MT, Sibug-Saber M, Cozen W, Liu L, Lynch CF, Wentzensen N, Jordan RC, Altekruse S, Anderson WF, Rosenberg PS, Gillison ML. Human papillomavirus and rising oropharyngeal cancer incidence in the United States. J Clin Oncol. 2011 Nov 10;29(32):4294-301. doi: 10.1200/JCO.2011.36.4596. Epub 2011 Oct 3. PMID 21969503
- [Background] Chaturvedi AK, Engels EA, Anderson WF, Gillison ML. Incidence trends for human papillomavirus-related and -unrelated oral squamous cell carcinomas in the United States. J Clin Oncol. 2008 Feb 1;26(4):612-9. doi: 10.1200/JCO.2007.14.1713. PMID 18235120
- [Background] Nasman A, Attner P, Hammarstedt L, Du J, Eriksson M, Giraud G, Ahrlund-Richter S, Marklund L, Romanitan M, Lindquist D, Ramqvist T, Lindholm J, Sparen P, Ye W, Dahlstrand H, Munck-Wikland E, Dalianis T. Incidence of human papillomavirus (HPV) positive tonsillar carcinoma in Stockholm, Sweden: an epidemic of viral-induced carcinoma? Int J Cancer. 2009 Jul 15;125(2):362-6. doi: 10.1002/ijc.24339. PMID 19330833
- [Background] Andl T, Kahn T, Pfuhl A, Nicola T, Erber R, Conradt C, Klein W, Helbig M, Dietz A, Weidauer H, Bosch FX. Etiological involvement of oncogenic human papillomavirus in tonsillar squamous cell carcinomas lacking retinoblastoma cell cycle control. Cancer Res. 1998 Jan 1;58(1):5-13. PMID 9426048
- [Background] Munger K, Baldwin A, Edwards KM, Hayakawa H, Nguyen CL, Owens M, Grace M, Huh K. Mechanisms of human papillomavirus-induced oncogenesis. J Virol. 2004 Nov;78(21):11451-60. doi: 10.1128/JVI.78.21.11451-11460.2004. No abstract available. PMID 15479788
- [Background] Psyrri A, DeFilippis RA, Edwards AP, Yates KE, Manuelidis L, DiMaio D. Role of the retinoblastoma pathway in senescence triggered by repression of the human papillomavirus E7 protein in cervical carcinoma cells. Cancer Res. 2004 May 1;64(9):3079-86. doi: 10.1158/0008-5472.can-03-3739. PMID 15126344
- [Background] Weinberger PM, Yu Z, Haffty BG, Kowalski D, Harigopal M, Brandsma J, Sasaki C, Joe J, Camp RL, Rimm DL, Psyrri A. Molecular classification identifies a subset of human papillomavirus--associated oropharyngeal cancers with favorable prognosis. J Clin Oncol. 2006 Feb 10;24(5):736-47. doi: 10.1200/JCO.2004.00.3335. Epub 2006 Jan 9. PMID 16401683
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Background] Gillison ML, Koch WM, Capone RB, Spafford M, Westra WH, Wu L, Zahurak ML, Daniel RW, Viglione M, Symer DE, Shah KV, Sidransky D. Evidence for a causal association between human papillomavirus and a subset of head and neck cancers. J Natl Cancer Inst. 2000 May 3;92(9):709-20. doi: 10.1093/jnci/92.9.709. PMID 10793107
- [Background] Gillison ML. Human papillomavirus and prognosis of oropharyngeal squamous cell carcinoma: implications for clinical research in head and neck cancers. J Clin Oncol. 2006 Dec 20;24(36):5623-5. doi: 10.1200/JCO.2006.07.1829. No abstract available. PMID 17179099
- [Background] Ringstrom E, Peters E, Hasegawa M, Posner M, Liu M, Kelsey KT. Human papillomavirus type 16 and squamous cell carcinoma of the head and neck. Clin Cancer Res. 2002 Oct;8(10):3187-92. PMID 12374687
- [Background] Lassen P, Eriksen JG, Hamilton-Dutoit S, Tramm T, Alsner J, Overgaard J. Effect of HPV-associated p16INK4A expression on response to radiotherapy and survival in squamous cell carcinoma of the head and neck. J Clin Oncol. 2009 Apr 20;27(12):1992-8. doi: 10.1200/JCO.2008.20.2853. Epub 2009 Mar 16. PMID 19289615
- [Background] Licitra L, Perrone F, Bossi P, Suardi S, Mariani L, Artusi R, Oggionni M, Rossini C, Cantu G, Squadrelli M, Quattrone P, Locati LD, Bergamini C, Olmi P, Pierotti MA, Pilotti S. High-risk human papillomavirus affects prognosis in patients with surgically treated oropharyngeal squamous cell carcinoma. J Clin Oncol. 2006 Dec 20;24(36):5630-6. doi: 10.1200/JCO.2005.04.6136. PMID 17179101
- [Background] Cmelak AJ, Li S, Goldwasser MA, Murphy B, Cannon M, Pinto H, Rosenthal DI, Gillison M, Forastiere AA. Phase II trial of chemoradiation for organ preservation in resectable stage III or IV squamous cell carcinomas of the larynx or oropharynx: results of Eastern Cooperative Oncology Group Study E2399. J Clin Oncol. 2007 Sep 1;25(25):3971-7. doi: 10.1200/JCO.2007.10.8951. PMID 17761982
- [Background] Fakhry C, Westra WH, Li S, Cmelak A, Ridge JA, Pinto H, Forastiere A, Gillison ML. Improved survival of patients with human papillomavirus-positive head and neck squamous cell carcinoma in a prospective clinical trial. J Natl Cancer Inst. 2008 Feb 20;100(4):261-9. doi: 10.1093/jnci/djn011. Epub 2008 Feb 12. PMID 18270337
- [Background] Worden FP, Kumar B, Lee JS, Wolf GT, Cordell KG, Taylor JM, Urba SG, Eisbruch A, Teknos TN, Chepeha DB, Prince ME, Tsien CI, D'Silva NJ, Yang K, Kurnit DM, Mason HL, Miller TH, Wallace NE, Bradford CR, Carey TE. Chemoselection as a strategy for organ preservation in advanced oropharynx cancer: response and survival positively associated with HPV16 copy number. J Clin Oncol. 2008 Jul 1;26(19):3138-46. doi: 10.1200/JCO.2007.12.7597. Epub 2008 May 12. PMID 18474879
- [Background] Rischin D, Young RJ, Fisher R, Fox SB, Le QT, Peters LJ, Solomon B, Choi J, O'Sullivan B, Kenny LM, McArthur GA. Prognostic significance of p16INK4A and human papillomavirus in patients with oropharyngeal cancer treated on TROG 02.02 phase III trial. J Clin Oncol. 2010 Sep 20;28(27):4142-8. doi: 10.1200/JCO.2010.29.2904. Epub 2010 Aug 9. PMID 20697079
- [Background] Lorch JH, Goloubeva O, Haddad RI, Cullen K, Sarlis N, Tishler R, Tan M, Fasciano J, Sammartino DE, Posner MR; TAX 324 Study Group. Induction chemotherapy with cisplatin and fluorouracil alone or in combination with docetaxel in locally advanced squamous-cell cancer of the head and neck: long-term results of the TAX 324 randomised phase 3 trial. Lancet Oncol. 2011 Feb;12(2):153-9. doi: 10.1016/S1470-2045(10)70279-5. Epub 2011 Jan 11. PMID 21233014
- [Background] Posner MR, Lorch JH, Goloubeva O, Tan M, Schumaker LM, Sarlis NJ, Haddad RI, Cullen KJ. Survival and human papillomavirus in oropharynx cancer in TAX 324: a subset analysis from an international phase III trial. Ann Oncol. 2011 May;22(5):1071-1077. doi: 10.1093/annonc/mdr006. Epub 2011 Feb 11. PMID 21317223
- [Background] Machtay M, Moughan J, Trotti A, Garden AS, Weber RS, Cooper JS, Forastiere A, Ang KK. Factors associated with severe late toxicity after concurrent chemoradiation for locally advanced head and neck cancer: an RTOG analysis. J Clin Oncol. 2008 Jul 20;26(21):3582-9. doi: 10.1200/JCO.2007.14.8841. Epub 2008 Jun 16. PMID 18559875
- [Background] Adelstein DJ, Li Y, Adams GL, Wagner H Jr, Kish JA, Ensley JF, Schuller DE, Forastiere AA. An intergroup phase III comparison of standard radiation therapy and two schedules of concurrent chemoradiotherapy in patients with unresectable squamous cell head and neck cancer. J Clin Oncol. 2003 Jan 1;21(1):92-8. doi: 10.1200/JCO.2003.01.008. PMID 12506176
- [Background] Forastiere A, Maor M, Weber R, Pajak, T, Glisson B, Trotti A, Ridge J, et al. Long term results of Intergroup RTOG 91-11: A Phase III trial to preserve the larynx - Induction cisplatin/5-FU and radiation therapy versus concurrent cisplatin and radiation therapy versus radiation therapy. Proceedings of the American Society of Clinical Oncology. 2006:5517.
- [Background] Staar S, Rudat V, Stuetzer H, Dietz A, Volling P, Schroeder M, Flentje M, Eckel HE, Mueller RP. Intensified hyperfractionated accelerated radiotherapy limits the additional benefit of simultaneous chemotherapy--results of a multicentric randomized German trial in advanced head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2001 Aug 1;50(5):1161-71. doi: 10.1016/s0360-3016(01)01544-9. PMID 11483325
- [Background] Taylor SG 4th, Murthy AK, Vannetzel JM, Colin P, Dray M, Caldarelli DD, Shott S, Vokes E, Showel JL, Hutchinson JC, et al. Randomized comparison of neoadjuvant cisplatin and fluorouracil infusion followed by radiation versus concomitant treatment in advanced head and neck cancer. J Clin Oncol. 1994 Feb;12(2):385-95. doi: 10.1200/JCO.1994.12.2.385. PMID 8113846
- [Background] Best SR, Ha PK, Blanco RG, Saunders JR Jr, Zinreich ES, Levine MA, Pai SI, Walker M, Trachta J, Ulmer K, Murakami P, Thompson R, Califano JA, Messing BP. Factors associated with pharyngoesophageal stricture in patients treated with concurrent chemotherapy and radiation therapy for oropharyngeal squamous cell carcinoma. Head Neck. 2011 Dec;33(12):1727-34. doi: 10.1002/hed.21657. Epub 2011 Jan 18. PMID 21246640
- [Background] Bonner JA, Harari PM, Giralt J, Cohen RB, Jones CU, Sur RK, Raben D, Baselga J, Spencer SA, Zhu J, Youssoufian H, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for locoregionally advanced head and neck cancer: 5-year survival data from a phase 3 randomised trial, and relation between cetuximab-induced rash and survival. Lancet Oncol. 2010 Jan;11(1):21-8. doi: 10.1016/S1470-2045(09)70311-0. Epub 2009 Nov 10. PMID 19897418
- [Background] Agoston ES, Robinson SJ, Mehra KK, Birch C, Semmel D, Mirkovic J, Haddad RI, Posner MR, Kindelberger D, Krane JF, Brodsky J, Crum CP. Polymerase chain reaction detection of HPV in squamous carcinoma of the oropharynx. Am J Clin Pathol. 2010 Jul;134(1):36-41. doi: 10.1309/AJCP1AAWXE5JJCLZ. PMID 20551264
- [Background] Harris SL, Thorne LB, Seaman WT, Hayes DN, Couch ME, Kimple RJ. Association of p16(INK4a) overexpression with improved outcomes in young patients with squamous cell cancers of the oral tongue. Head Neck. 2011 Nov;33(11):1622-7. doi: 10.1002/hed.21650. Epub 2010 Dec 28. PMID 21990227
- [Background] Schache AG, Liloglou T, Risk JM, Filia A, Jones TM, Sheard J, Woolgar JA, Helliwell TR, Triantafyllou A, Robinson M, Sloan P, Harvey-Woodworth C, Sisson D, Shaw RJ. Evaluation of human papilloma virus diagnostic testing in oropharyngeal squamous cell carcinoma: sensitivity, specificity, and prognostic discrimination. Clin Cancer Res. 2011 Oct 1;17(19):6262-71. doi: 10.1158/1078-0432.CCR-11-0388. PMID 21969383
- [Background] Maxwell JH, Kumar B, Feng FY, Worden FP, Lee JS, Eisbruch A, Wolf GT, Prince ME, Moyer JS, Teknos TN, Chepeha DB, McHugh JB, Urba SG, Stoerker J, Walline HM, Kurnit DM, Cordell KG, Davis SJ, Ward PD, Bradford CR, Carey TE. Tobacco use in human papillomavirus-positive advanced oropharynx cancer patients related to increased risk of distant metastases and tumor recurrence. Clin Cancer Res. 2010 Feb 15;16(4):1226-35. doi: 10.1158/1078-0432.CCR-09-2350. Epub 2010 Feb 9. PMID 20145161
- [Background] Anderson KS, Wong J, D'Souza G, Riemer AB, Lorch J, Haddad R, Pai SI, Longtine J, McClean M, LaBaer J, Kelsey KT, Posner M. Serum antibodies to the HPV16 proteome as biomarkers for head and neck cancer. Br J Cancer. 2011 Jun 7;104(12):1896-905. doi: 10.1038/bjc.2011.171. PMID 21654689
- [Background] Kumar B, Cordell KG, Lee JS, Worden FP, Prince ME, Tran HH, Wolf GT, Urba SG, Chepeha DB, Teknos TN, Eisbruch A, Tsien CI, Taylor JM, D'Silva NJ, Yang K, Kurnit DM, Bauer JA, Bradford CR, Carey TE. EGFR, p16, HPV Titer, Bcl-xL and p53, sex, and smoking as indicators of response to therapy and survival in oropharyngeal cancer. J Clin Oncol. 2008 Jul 1;26(19):3128-37. doi: 10.1200/JCO.2007.12.7662. Epub 2008 May 12. PMID 18474878
- [Background] Porceddu SV, Pryor DI, Burmeister E, Burmeister BH, Poulsen MG, Foote MC, Panizza B, Coman S, McFarlane D, Coman W. Results of a prospective study of positron emission tomography-directed management of residual nodal abnormalities in node-positive head and neck cancer after definitive radiotherapy with or without systemic therapy. Head Neck. 2011 Dec;33(12):1675-82. doi: 10.1002/hed.21655. Epub 2011 Jan 14. PMID 22076976
- [Background] Riemer AB, Keskin DB, Zhang G, Handley M, Anderson KS, Brusic V, Reinhold B, Reinherz EL. A conserved E7-derived cytotoxic T lymphocyte epitope expressed on human papillomavirus 16-transformed HLA-A2+ epithelial cancers. J Biol Chem. 2010 Sep 17;285(38):29608-22. doi: 10.1074/jbc.M110.126722. Epub 2010 Jul 8. PMID 20615877
- [Background] Misiukiewicz K, Gupta V, Miles BA, Bakst R, Genden E, Selkridge I, Surgeon JT, Rainey H, Camille N, Roy E, Zhang D, Ye F, Jia R, Moshier E, Bonomi M, Hwang M, Som P, Posner MR. Standard of care vs reduced-dose chemoradiation after induction chemotherapy in HPV+ oropharyngeal carcinoma patients: The Quarterback trial. Oral Oncol. 2019 Aug;95:170-177. doi: 10.1016/j.oraloncology.2019.06.021. Epub 2019 Jun 25. PMID 31345387

DOCUMENTS (1):
  • Informed Consent Form (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT02945631/ICF_000.pdf